CLINICAL TRIAL: NCT04863599
Title: Patient Experience With OMS Procedures Under General Anesthesia Compared to Sedation
Brief Title: Patient Experience With OMS Procedures Regarding Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Dieter Mesotten, MD, Ziekenhuis Oost-Limburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Z-2021038
Record Dates: First submitted 2021-04-26; First posted 2021-04-28 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Patient Satisfaction
Keywords: General anesthesia; Sedation
MeSH Terms: conditions — Patient Satisfaction | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OMS procedure under general anesthesia or sedation (Other): Questionnaire
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Patients will be asked to complete the Bauer and Brice questionnaire at post-operative day 1.

SUMMARY:
The main purpose of the study is to know more about the experience/satisfaction of patients undergoing oral and maxillofacial surgery (OMS). Depending on the type of procedure, the patient will receive a sedation or a general anesthesia. At the first day post-operatively, patients will be contacted to complete a questionnaire. The questionnaire will be subdivided into anaesthesia-related discomfort and anaesthesia care in general.

ELIGIBILITY:
Inclusion Criteria:

* OMS procedure
* signed informed consent
* Age above 12 years

Exclusion Criteria:

* need for post-operative hospitalization
* mental disorder with no capability of filling in questionnaires

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2021-09-21 (Actual)

PRIMARY OUTCOMES:
Bauer questionnaire at post-operative day 1 | post-operative day 1
  The Bauer questionnaire contains a set of questions on anaesthesia-related discomfort and another set on satisfaction with anaesthesia care in general. The questions on discomfort will be assessed on a 3-point scale, and those on patient satisfaction on a 4-point scale.
Brice questionnaire at post-operative day 1 | post-operative day 1
  The questionnaire attempts to identify patients who may have had memories of their operation i.e. accidental awareness under anesthesia. These are open questions.

CONTACTS AND LOCATIONS:
Overall Officials: Joris Vundelinckx, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium

IPD SHARING:
Plan to Share IPD: No